CLINICAL TRIAL: NCT05728671
Title: An Open-Label, Bioavailability Study to Compare Liquid vs Two Solid Formulations of IP2015 in Healthy Male Subjects
Brief Title: Bioavailability Study to Compare Liquid vs Two Solid Formulations of IP2015
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Initiator Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IP2015CS04
Record Dates: First submitted 2022-12-20; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2022-12

CONDITIONS: Bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IP2015_PO release form 1 (Experimental): Test formulation 1
  Interventions: Drug: IP2015
- IP2015_PO release form 2 (Experimental): Test formulation 2
  Interventions: Drug: IP2015
- IP2015_PO release form 3 (Experimental): Test formulation 3
  Interventions: Drug: IP2015

INTERVENTIONS:
Drug: IP2015 — Test drug

SUMMARY:
The study's primary objective is to determine the bioavailability of two solid formulations of IP2015 compared to a liquid formulation of IP2015 in healthy male subjects

DETAILED DESCRIPTION:
It is planned to include 12 subjects. Each subject will take part in three treatment periods, in which they will receive a single dose of IP2015 liquid and then to different IP2015 solid formulations, respectively, in each treatment period. Overall, each subject will receive each treatment once only.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) of 18 to 30 kg/m2, inclusive.
* Subject is ≥50 kg.
* Healthy as determined by a responsible physician, based on medical evaluation including medical history, physical examination, concomitant medication, vital signs, 12-lead ECG, clinical laboratory evaluations.

Exclusion Criteria:

* Any significant CNS, cardiac, pulmonary, metabolic, renal, hepatic (including Gilbert's syndrome), gastrointestinal (GI) or psychiatric conditions, or history of fainting or syncope or such condition that, in the opinion of the Investigator, may place the subject at an unacceptable risk as a participant in the study, may interfere with the interpretation of safety or tolerability data obtained in this study, or may interfere with the absorption, distribution, metabolism or excretion (ADME) of drugs, or with the completion of treatment according to this Protocol.
* Clinically relevant history of abnormal physical or mental health interfering with the study as determined by medical history and physical examinations obtained during Screening as judged by the Investigator (including [but not limited to], neurological, psychiatric, endocrine, cardiovascular, respiratory, GI, hepatic or renal disorder).
* Clinically relevant abnormal laboratory results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis), 12-lead ECG and vital signs or physical findings at Screening. In case of uncertain or questionable results, tests performed during Screening may be repeated to confirm eligibility or judged to be clinically irrelevant for healthy subjects.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2023-02-16 (Estimated); Primary Completion 2023-05-16 (Estimated); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
AUC | 72 hours
  Pharmacokinetics
Tmax | 72 hours
  Pharmacokinetics
Cmax | 72 hours
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Connell, MD, Principal Investigator — MAC UK

IPD SHARING:
Plan to Share IPD: No